CLINICAL TRIAL: NCT01645826
Title: Calcium Channel Blockers in Nitric Oxide Non-responder Pulmonary Arterial Hypertension.
Brief Title: Efficacy Study of Cardizem in Pulmonary Arterial Hypertension
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants agreed to enroll since study start
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Mark Rumbak, Professor of Medicine, Internal Medicine, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00004379
Record Dates: First submitted 2011-10-18; First posted 2012-07-20 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Idiopathic Pulmonary Arterial Hypertension; Primary Pulmonary Hypertension; Pulmonary Arterial Hypertension; Familial Primary Pulmonary Hypertension
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension; Pulmonary Arterial Hypertension | interventions — Diltiazem; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diltiazem (Experimental): The study agent will be Diltiazem and will start at 60 mg po BID then titrated up every two weeks until at a maximum dose of 180mg po BID.
  Interventions: Drug: Diltiazem Hydrochloride
- Sugar Pill (Placebo Comparator): The placebo group of patients will be treated with Drug A (sugar pill) PO bid and titrated up every two weeks for next titration dose (actually will be an unchanged concentration).
  Interventions: Drug: Sugar Pill

INTERVENTIONS:
Drug: Diltiazem Hydrochloride — The study agent will be diltiazem and will start at 60 mg po BID then titrated up very two weeks until at a maximum maintenance dose of 180mg po BID for six weeks.
  Other Names: cardizem; treatment group
  Arms: Diltiazem
Drug: Sugar Pill — The placebo group of patients will be treated with sugar pill PO bid and return every two weeks for next titration dose (actually will be an unchanged concentration).
  Other Names: placebo
  Arms: Sugar Pill

SUMMARY:
The purpose of this study is to determine if cardizem is effective in the treatment of nitric oxide non-responder pulmonary arterial hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants
* Confirmed WHO class I pulmonary arterial hypertension
* Nitric Oxide Non-Responders on right heart catheterization
* Experience dyspnea, NYHA III-IV with poor oxygenation and quality of life despite standard treatments
* Must be able to swallow medications

Exclusion Criteria:

* Pulmonary hypertension secondary to 1) elevations in pulmonary venous pressures (i.e. left heart disease), 2) chronic hypoxemic states from lung diseases such as COPD, sleep-disordered breathing, alveolar hypoventilation disorders, chronic exposure to high altitude and developmental abnormalities 3) chronic thromboembolic disease, 4) sarcoidosis, 5) Lymphangiomyomatosis, 5) Pulmonary Langerhans Cell Histiocytosis
* Already on a calcium channel blocker
* Systolic blood pressure less than 90
* Heart rate less than 55
* Pregnant
* Cannot sign informed consent
* Right heart failure
* Pulmonary Veno-occlusive disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Six Minute Walk Distance | 12 weeks

SECONDARY OUTCOMES:
Dyspnea Score | 12 weeks
Quality of Life Score | 12 weeks
Pulse Oximetry | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rumbak, MD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

REFERENCES:
- [Background] Badesch DB, Abman SH, Simonneau G, Rubin LJ, McLaughlin VV. Medical therapy for pulmonary arterial hypertension: updated ACCP evidence-based clinical practice guidelines. Chest. 2007 Jun;131(6):1917-28. doi: 10.1378/chest.06-2674. PMID 17565025
- [Background] Aromatorio GJ, Uretsky BF, Reddy PS. Hypotension and sinus arrest with nifedipine in pulmonary hypertension. Chest. 1985 Feb;87(2):265-7. doi: 10.1378/chest.87.2.265. PMID 3967536
- [Background] Batra AK, Segall PH, Ahmed T. Pulmonary edema with nifedipine in primary pulmonary hypertension. Respiration. 1985;47(3):161-3. doi: 10.1159/000194763. PMID 4001571
- [Background] Chaouat A, Kessler R, Weitzenblum E. Pulmonary oedema and pleural effusion in two patients with primary pulmonary hypertension treated with calcium channel blockers. Heart. 1996 Apr;75(4):383. doi: 10.1136/hrt.75.4.383. No abstract available. PMID 8705766
- [Background] Clarke WR, Horn JR, Kawabori I, Gurtel S. Potentially serious drug interactions secondary to high-dose diltiazem used in the treatment of pulmonary hypertension. Pharmacotherapy. 1993 Jul-Aug;13(4):402-5. PMID 8361869
- [Background] Farber HW, Karlinsky JB, Faling LJ. Fatal outcome following nifedipine for pulmonary hypertension. Chest. 1983 Apr;83(4):708-9. doi: 10.1378/chest.83.4.708. No abstract available. PMID 6831965
- [Background] Holcomb BW Jr, Loyd JE, Ely EW, Johnson J, Robbins IM. Pulmonary veno-occlusive disease: a case series and new observations. Chest. 2000 Dec;118(6):1671-9. PMID 11115457
- [Background] Houtchens J, Martin D, Klinger JR. Diagnosis and management of pulmonary arterial hypertension. Pulm Med. 2011;2011:845864. doi: 10.1155/2011/845864. Epub 2011 Sep 20. PMID 21941650
- [Background] Nauser TD, Stites SW. Diagnosis and treatment of pulmonary hypertension. Am Fam Physician. 2001 May 1;63(9):1789-98. PMID 11352291
- [Background] McLaughlin VV, Archer SL, Badesch DB, Barst RJ, Farber HW, Lindner JR, Mathier MA, McGoon MD, Park MH, Rosenson RS, Rubin LJ, Tapson VF, Varga J; American College of Cardiology Foundation Task Force on Expert Consensus Documents; American Heart Association; American College of Chest Physicians; American Thoracic Society, Inc; Pulmonary Hypertension Association. ACCF/AHA 2009 expert consensus document on pulmonary hypertension a report of the American College of Cardiology Foundation Task Force on Expert Consensus Documents and the American Heart Association developed in collaboration with the American College of Chest Physicians; American Thoracic Society, Inc.; and the Pulmonary Hypertension Association. J Am Coll Cardiol. 2009 Apr 28;53(17):1573-619. doi: 10.1016/j.jacc.2009.01.004. No abstract available. PMID 19389575
- [Background] Galie N, Torbicki A, Barst R, Dartevelle P, Haworth S, Higenbottam T, Olschewski H, Peacock A, Pietra G, Rubin LJ, Simonneau G, Priori SG, Garcia MA, Blanc JJ, Budaj A, Cowie M, Dean V, Deckers J, Burgos EF, Lekakis J, Lindahl B, Mazzotta G, McGregor K, Morais J, Oto A, Smiseth OA, Barbera JA, Gibbs S, Hoeper M, Humbert M, Naeije R, Pepke-Zaba J; Task Force. Guidelines on diagnosis and treatment of pulmonary arterial hypertension. The Task Force on Diagnosis and Treatment of Pulmonary Arterial Hypertension of the European Society of Cardiology. Eur Heart J. 2004 Dec;25(24):2243-78. doi: 10.1016/j.ehj.2004.09.014. No abstract available. PMID 15589643
- See also: Robbins, Ivan. The Role of Calcium Channel Blockers in Pulmonary Arterial Hypertension. 2006 Feb 23. — http://www.medscape.org/viewarticle/523338